CLINICAL TRIAL: NCT02541760
Title: Monteleukast Versus Inhaled Mometasone for Treatment of Otitis Media With Effusion in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Principal Investigator, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 163
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Otitis Media With Effiusion
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Montelukast (Experimental): 4 ml monteleukast daily for one month
  Interventions: Drug: Monteleukast
- Mometasone (Active Comparator): Inhaled mometasone 1 puff in each side of nose for one month
  Interventions: Drug: Mometasone
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Monteleukast — 4 ml monteleukast daily for one month
  Arms: Montelukast
Drug: Mometasone — Inhaled mometasone 1 puff in each side of nose for one month
  Arms: Mometasone

SUMMARY:
Otitis media is one of the most common infections among children and is a complication in about 30% of common colds. The most common complication of acute otitis media is otitis media with effusion. Some studies have reported the effects of montelukast and mometasone nasal spray in treatment of otitis media with effusion. However, current information is inadequate in this issue. The aim of this study was to compare the effectiveness of montelukast and mometasone nasal spray in treatment of otitis media with effusion in children attending Koodakan hospital in Bandar Abbas, Iran.

ELIGIBILITY:
Inclusion Criteria:

* • Children who were between 2 to 6 years old

  * Definite diagnosis of OME with symptoms and examination

Exclusion Criteria:

* • Currently were using corticosteroids or prophylactic monteleukast

  * Chronic pulmonary or cardiac diseases or immune deficiency
  * Allergic rhinitis
  * Hypersensitivity to monteleukast or corticosteroids
  * Avoidance of parents to fill the written informed consent

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Treatment response | 1 months
  Defined as complete, partial, or no response based on the physician examination

SECONDARY OUTCOMES:
Drug side effects | 1 month
  Frequency of Drug side effects as reported by the children or their parents

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Mahboobi, M.D, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran

REFERENCES:
- [Derived] Mulvaney CA, Galbraith K, Webster KE, Rana M, Connolly R, Tudor-Green B, Marom T, Daniel M, Venekamp RP, Schilder AG, MacKeith S. Topical and oral steroids for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Dec 13;12(12):CD015255. doi: 10.1002/14651858.CD015255.pub2. PMID 38088821
- [Derived] Rahmati MB, Safdarian F, Shiroui B, Zare S, Sadeghi N. Montelukast versus inhaled mometasone for treatment of otitis media with effusion in children: A randomized controlled trial. Electron Physician. 2017 Jul 25;9(7):4890-4894. doi: 10.19082/4890. eCollection 2017 Jul. PMID 28894551